CLINICAL TRIAL: NCT05913947
Title: Lithium Versus Cariprazine in the Acute Phase Treatment of Bipolar Depression: a Pragmatic Head-to-head Open, Randomized Multicenter Study: The 9th Study of the Danish University Antidepressant Group (DUAG 9)
Brief Title: Lithium Versus Cariprazine in the Acute Phase Treatment of Bipolar Depression (DUAG9)
Acronym: DUAG9
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Mental Health Department Odense, University Clinic (Unknown); Psychiatric Center Copenhagen, Rigshospitalet (Unknown); Psychiatric Hospital, Hillerod (Other)
Responsible Party: Principal Investigator, René Ernst Nielsen, MD, PhD, Professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-006706-69
Record Dates: First submitted 2023-03-29; First posted 2023-06-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; lithium citrate; cariprazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium (Experimental): Lithium citrate from 12 mmol increased to result in af 12-hour se-lithium between 0.6 and 0.8 mmol/l
  Interventions: Drug: Lithium
- Cariprazine (Experimental): Cariprazine from 1.5 mg to 3 mg daily in a single dose.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Lithium — The starting dose (day one) of lithium citrate is 12 mmol (one tablet of lithium citrate contains 6 mmol lithium) given once a day before bedtime. On day three the dose is increased to 18 mmol. Dose adjustments are permitted after 7 days in a flexible manner to result in a 12-hour se-lithium between 0.6 and 0.8 mmol/l, aiming for the upper limit at the treating physician's discretion.
  Other Names: Litarex, ATC; N05AN01
  Arms: Lithium
Drug: Cariprazine — The starting dose for cariprazine is 1.5 mg daily in a single dose, and subsequently, after a minimum of two weeks, the dose can be increased to 3 mg and decreased again to 1.5 mg daily at the treating physician's discretion.
  Other Names: Reagila, ATC: N05AX15
  Arms: Cariprazine

SUMMARY:
The goal is to study the effect of lithium compared to cariprazine in patients with depression in a bipolar disease.

The main question it aims to answer is:

Difference in change between the two groups from baseline to after 8 weeks treatment on Hamilton Ratings Scale for Depression, 6-item version (HDS-6)

Participants will be randomized to treatment with either lithium or cariprazin.

* Will meet for interview and ratings 4 times during study period.
* In two meetings, there will be made blood samples and ECG. At one meeting also a Urine sample.
* Will be contacted for telephone interviews at 6 occasions.

DETAILED DESCRIPTION:
The primary aim is to investigate whether cariprazine is superior to lithium or vice versa in the acute treatment of patients with bipolar type 1 or 2 in a current depressive episode measured as change on the Hamilton Depression Scale, 6 item version (HDS-6) from baseline to 8 weeks of treatment. Secondarily, we aimed at comparing the two study medications on various other clinically relevant variables.

These include depressive and manic symptomatology, sleep patterns, general well-being, cognitive function, social functioning and suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of bipolar disorder, type 1 or type 2, and a current episode of depression according to DSM-5
* Severity of depression: A score of at least 21 on the self-reported Major Depression Inventory (MDI).
* No start or dose increase of psychotropic medication (except for benzodiazepines and benzodiazepine-like drugs (zopiclone, zolpidem, and melatonin)) in the two weeks prior to inclusion.
* No new start of formalized psychotherapy sessions, excluding psychoeducation, during the 4 weeks prior to inclusion.
* Age criteria: Subjects must be at least 18 years old and below 65 at the time of randomization.
* The duration of the current depressive episode must be between 4 and 52 weeks as judged by the investigator at the time of randomization.
* Clinical uncertainty regarding which of the alternatives, cariprazine and lithium, would be the better choice in the specific case.
* Female participants should be sterile or non-fertile or, in case of being fertile, they must have a negative pregnancy test AND use safe anticonception.
* Signed document of informed consent.

Exclusion Criteria:

* Prior or ongoing acute treatment of a depressive episode lasting > 14 days with either lithium or cariprazine as judged by the investigator.
* ECT within the current depressive episode.
* A score of MAS > 6.
* A diagnosis of dementia.
* High risk of non-adherence at the investigator's discretion.
* Not understanding the Danish language as judged by the investigator
* Psychiatric coercion in the form of forced admission or detainment OR sentence to forensic psychiatric care.
* Presence of clinically relevant delusions, hallucinations or other psychotic symptoms as judged by the investigator.
* Suicidality according to C-SSRS with a positive response to question 4 or 5 or upon investigator's discretion.
* Medical conditions like cancer, kidney failure, epilepsy, deep brain stimulation device, or other medical conditions interfering with study the outcome and safety as judged by investigator's discretion.
* Current harmful use or dependency of alcohol or drugs according to DSM-5.
* Known allergy to any of the substances in the study medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-02 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depressions scale, version 6 (HDS-6) | 8 weeks
  The primary aim is to investigate whether cariprazine is superior to lithium or vice versa in the acute treatment of patients with bipolar type 1 or 2 in a current depressive episode measured as change on the Hamilton Depression Scale, 6 item version, HDS-6. (Values 0- 22, higher scores mean a worse outcome).

SECONDARY OUTCOMES:
Difference-in-difference for HDS-17 | Week 4 and 8
  Difference-in-differences for secondary continuous measures: Hamilton Depression Scale, 17 item version, HDS-17. (Values 0- 52, higher scores mean a worse outcome)
Difference-in-differences in HDS-6 for the PP 8 population | 8 weeks
  Difference-in-differences (baseline to 8 weeks) in HDS-6 for the PP 8 population.
  Hamilton Depression Scale, 6 item version, HDS-6. (Values 0- 22, higher scores mean a worse outcome).
Between-groups difference in proportion of responders and remitters in HDS-6 Scores. | Week 4 and week 8
  Between-groups difference in proportion of responders and remitters at week 4 and 8 in HDS-6 scores.
  Hamilton Depression Scale, 6 item version, HDS-6. (Values 0- 22, higher scores mean a worse outcome).
Between-groups difference in proportion of responders and remitters | Week 4 and 8
  Between-groups difference in proportion of responders and remitters with response and remission defined by HDS-6 score without clinical relevant manic symptoms (MAS <7) at planned or premature endpoint.
  Hamilton Depression Scale, 6 item version, HDS-6. (Values 0- 22, higher scores mean a worse outcome).
Between-groups difference in the proportion of patients with 'acceptable wellbeing' | up to 8 weeks
  Between-groups difference in the proportion of patients with 'acceptable wellbeing', defined as the subject reporting ≥50 on the WHO-5 questionnaire at endpoint. WHO-five Well-being Index, WHO-5 (Values 0- 100, higher scores mean a better outcome).
Between-groups difference in proportion of switches to mania/hypomania. | up to 8 weeks
  Between-groups difference in proportion of switches to mania/hypomania with or without mixed features, defined as mania/hypomania after DSM-5 or symptoms requiring treatment (switch or response occurring at any time in the study period)
Between-groups difference in "(switch to mania or hypomania) / (response) -ratio", | up to 8 weeks
  Between-groups difference in "(switch to mania or hypomania) / (response) -ratio", defined as the number of subjects switching to mania or hypomania (as defined above) divided by the total number of responders, including those responders switching to mania
Between-group differences in reason for and time to all cause treatment discontinuation | up to 8 weeks
  Between-group differences in reason for and time to all cause treatment discontinuation (lack of effect, lack of tolerability, lost to follow-up, or other cause).
Between-group difference in treatment compliance. | up to 8 weeks
  Between-group difference in treatment compliance. Treatment compliance is defined as the proportion of received treatments out of the planned until drop-out or end of study.
Between-group difference in reasons for premature discontinuation | up to 8 weeks
  Between-group difference for the ITT population in reasons for premature discontinuation
Difference-in-difference for MAS | Week 4 and 8
  Difference-in-differences for secondary continuous measures: MAS Bech-Rafaelsens Mania scale .(Values 0- 44, higher scores mean a worse outcome).
Difference-in-difference for MES | Week 4 and 8
  Difference-in-differences for secondary continuous measures: MES Bech-Rafaelsens Melancholia scale, MES .(Values 0- 44, higher scores mean a worse outcome).
Difference-in-differences for MADRS | Week 4 and 8
  Difference-in-differences for secondary continuous measures: MADRS Montgomery-Aaberg Depression Rating Scale, MADRS .(Values 0- 60, higher scores mean a worse outcome).
Difference-in-difference for YMRS | Week 4 and 8
  Difference-in-differences for secondary continuous measures:YMRS Young Mania Rating Scale, YMRS .(Values 0- 60, higher scores mean a worse outcome).
Difference-in-differences for ASRM-14 | Week 4 and 8
  Difference-in-differences for secondary continuous measures:ASRM-14 Altman Self-Rating Mania Scale-14, .(Values 0- 56, higher scores mean a worse outcome).
Difference-in-differences for MDI | Week 4 and 8
  Difference-in-differences for secondary continuous measures:MDI Major Depression Inventory, MDI (Values 0- 58, higher scores mean a worse outcome).
Difference-in-differences for WHO-5 questionnaire | Week 4 and 8
  Difference-in-differences for secondary continuous measures: WHO-5 questionnaire.
  WHO-five Well-beeing Index, WHO-5 (Values 0- 100, higher scores mean a better outcome).
Difference-in-difference for SCIP | Week 8
  Difference-in-differences for secondary continuous measures: SCIP Screen for Cognitive Impairment in Psychiatry, SCIP (Values 0- 64+, higher scores mean a better outcome)
Difference-in-difference for COBRA | Week 8
  Difference-in-differences for secondary continuous measures: COBRA Cognitive complaints in bipolar disorder Ratings assessment, COBRA, (Values 0- 48, higher scores mean a worse outcome).
Difference-in-difference for FAST | Week 4 and 8
  Difference-in-differences for secondary continuous measures: FAST Functioning Assessment Short Test, FAST (Values 0 - 72, higher scores mean a worse outcome).
Difference-in-difference for PSQI | Week 4 and 8
  Difference-in-differences for secondary continuous measures:PSQI PIttsburgh Sleep Quality Index, PSQI (Values 0 - 21, higher scores mean a worse outcome).
Difference-in-difference for CGI-S | Week 4 and 8
  Difference-in-differences for secondary continuous measures: CGI-S Clinical Global Impression Scale - Severity, CGI-S (Values 1 -7, higher scores mean a worse outcome).
Difference-in-difference for CGI-I | Week 4 and 8
  Difference-in-differences for secondary continuous measures:CGI-I Clinical Global Impression Scale - Global Improvement CGI- I (Values 1 -7, higher scores mean a worse outcome).
Difference-in-difference for C-SSRS | Week 4 and 8
  Difference-in-differences for secondary continuous measures: C-SSRS Columbia-Suicide Severity Rating Scale, C-SSRS (Values 1 - 5, higher scores mean a worse outcome).
Difference-in-difference for accumulated benzodiazepine dose | Up to 8 weeks
  Difference-in-differences for secondary continuous measures: accumulated benzodiazepine dose as diazepam equivalents (DSKP)
Difference-in-difference for time to all-causes discontinuation | Up to 8 weeks
  Difference-in-differences for secondary continuous measures: for time to all-causes discontinuation
Difference-in-difference for time to all-causes. all-causes study endpoint. | Up to 8 weeks
  Difference-in-differences for secondary continuous measures: all-causes study endpoint.
Between-group difference in reasons for time to all cause discontinuation. | Up to 8 weeks
  Between-group difference for the ITT population in reasons for time to all cause discontinuation.
Between-group difference in reasons for treatment expectation. | Up to 8 weeks
  Between-group difference for the ITT population in reasons for treatment expectation.
Between-group difference in reasons for adverse events. | Up to 8 weeks
  Between-group difference for the ITT population in reasons for adverse events.
Between-group difference in reasons for serious adverse events. | Up to 8 weeks
  Between-group difference for the ITT population in reasons for serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: René E. Nielsen, Prof, MD,PhD, Principal Investigator — Psychiatry, Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hovgesen SV, Licht RWW, Straszek SPV, Christensen AE, Vinberg M, Videbech P, Miskowiak KW, Johnsen S, Munk MM, Mai ML, Baethge C, Kessing LV, Nielsen RE. Lithium versus cariprazine in the acute phase treatment for depressive episodes in patients with bipolar disorder: a protocol for a pragmatic open, randomised multicentre study - the 9th trial of the Danish University Antidepressant Group, DUAG-9. BMJ Open. 2025 Aug 27;15(8):e102406. doi: 10.1136/bmjopen-2025-102406. PMID 40866064